CLINICAL TRIAL: NCT02493192
Title: Birth Ball Versus Meperidine and Haloperidol Injection for Pain Relief During First Stage of Labour
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Julia Fernandez, Julita Fernández Arranz, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V03_020911
Record Dates: First submitted 2015-06-23; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Parturition; Humanizing Deliver; Labor Pain; Natural Childbirth; Labor Onset; First Labor Stage
Keywords: Parturition; Humanizing Deliver; Labor Pain; Natural Childbirth; Labor Onset; First Labor Stage; Birth ball; meperidine; pethidine
MeSH Terms: conditions — Labor Pain | interventions — Meperidine; Haloperidol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meperidine (Active Comparator): Use pethidine and haloperidol injection as a pain relief.
  Interventions: Drug: pethidine and haloperidol injection
- birth ball (Experimental): Use birth ball as a pain relief.
  Interventions: Other: birth ball

INTERVENTIONS:
Drug: pethidine and haloperidol injection
  Other Names: meperidine and haloperidol injection
  Arms: Meperidine
Other: birth ball
  Other Names: fit ball, swiss ball
  Arms: birth ball

SUMMARY:
The study was performed at Gregorio Marañón Hospital birth centre. A Randomised Clinical Trial comparing the two methods of pain relief in the first time of labour was carried out. In this study, 110 women in the first stage of labour were allocated in two study groups by a randomised block design. One of them used the birth ball as a pain relief method,and the other one used pethidine and haloperidol injection.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* women in the first stage of labour or women at induction of labour
* fetal head in pelvis or whole amniotic membranes
* must be able to understand spanish

Exclusion Criteria:

* intrapartum meconium
* needed of continuous fetal monitoring
* suspecte/compromise fetal wellbeing
* morbidly obese women
* unaccompanied women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
pain | 24 months
  We use a numeric scale, since 0 ( no pain) to 10 (the greatest pain), to measure this item. We use it with women in the first stage of labour, with labor pain

SECONDARY OUTCOMES:
Baby´s apgar | 24 months
  We use the apgar Test to measure this item. Since 0 to 10.We use it after birth, with babies of women who are in our study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Gregorio Marañón, Madrid, Madrid, Spain

REFERENCES:
- [Background] Leung RW, Li JF, Leung MK, Fung BK, Fung LC, Tai SM, Sing C, Leung WC. Efficacy of birth ball exercises on labour pain management. Hong Kong Med J. 2013 Oct;19(5):393-9. doi: 10.12809/hkmj133921. Epub 2013 Jul 22. PMID 23878201
- [Background] Schult TM, Awosika ER, Schmunk SK, Hodgson MJ, Heymach BL, Parker CD. Sitting on stability balls: biomechanics evaluation in a workplace setting. J Occup Environ Hyg. 2013;10(2):55-63. doi: 10.1080/15459624.2012.748324. PMID 23252582
- [Background] Delgado-Garcia BE, Orts-Cortes MI, Poveda-Bernabeu A, Caballero-Perez P. [Randomised controlled clinical trial to determine the effects of the use of birth balls during labour]. Enferm Clin. 2012 Jan-Feb;22(1):35-40. doi: 10.1016/j.enfcli.2011.07.001. Epub 2011 Aug 31. Spanish. PMID 21885314
- [Background] Gau ML, Chang CY, Tian SH, Lin KC. Effects of birth ball exercise on pain and self-efficacy during childbirth: a randomised controlled trial in Taiwan. Midwifery. 2011 Dec;27(6):e293-300. doi: 10.1016/j.midw.2011.02.004. Epub 2011 Apr 3. PMID 21459499
- [Background] Taavoni S, Abdolahian S, Haghani H, Neysani L. Effect of birth ball usage on pain in the active phase of labor: a randomized controlled trial. J Midwifery Womens Health. 2011 Mar-Apr;56(2):137-40. doi: 10.1111/j.1542-2011.2010.00013.x. Epub 2011 Feb 28. PMID 21429078